CLINICAL TRIAL: NCT03355937
Title: The Effects of Using Microfluidic Separation Sperm Selection for Unexplained Infertility(UEI) and Reccurrent Implantation Failure(RIF)
Brief Title: Using Microfluidic Separation Sperm Selection for Unexplained Infertility and Reccurrent Implantation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Murat Dogan, Principal İnvestigator, Acibadem University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: Ob&Gyn Fulya
Record Dates: First submitted 2017-11-15; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Unexplained Infertility; Recurrent Implantation Failure
Keywords: unexplained infertility; recurrent implantation failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UEI Sperm Chip (-) (Active Comparator): Conventional IVF treatment and using conventional sperm selection
  Interventions: Procedure: Sperm Chip
- UEI Sperm Chip (+) (Experimental): Conventional IVF treatment and using sperm chip for sperm selection
  Interventions: Procedure: Sperm Chip
- RIF sperm chip (-) (Active Comparator): Conventional IVF treatment and using conventional sperm selection
  Interventions: Procedure: Sperm Chip
- RIF sperm chip (+) (Experimental): Conventional IVF treatment and using sperm chip for sperm selection
  Interventions: Procedure: Sperm Chip

INTERVENTIONS:
Procedure: Sperm Chip — Sperm selection using by conventional or with sperm chip

SUMMARY:
In order to increase the likelihood of achieving IVF-treated pregnancy, good quality embryo transfer is important. To get good quality embryos, good quality gametes are needed. The selection of sperm is regulated according to the changing and mobility characteristics of today's conditions. The choice of multi-fluid sperm is thought to provide better sperm to obtain the environment in physiological conditions. Better embryo transfer to achieve better sperm elongation will increase the likelihood of pregnancy.

DETAILED DESCRIPTION:
Patients will be treated with conventional IVF treatment. A vaginal ultrasound (US) examination will be perform on day 3 of the cycle for assessment of ovarian size and to exclude patients with large ovarian cysts. If a cyst >20 mm is present, the cycle will cancel. At an initial dose of 225 IU, hMG will be given daily by IM injection commencing on day 3 of the cycle. The dose will be adjusted as re- quired depending on the E2 (estradiol) level. Daily endovaginal US examinations for follicle growth assessment will be started when the E2 level reached 275 pg/mL (1,000 pmoljL). When at least two follicles would reach 18 mm in diameter, 5,000 IU of hCG will be administered intramuscularly. Oocyte retrieval will be performed vaginally under US guidance 36 hours later. Sperm for ICSI procedure of oocytes will be prepared by a standard swim-up technique using for control group and sperm chip method will be used for study group for Unexplained Infertility and Recurrent Implantation Failure group. Uterine transfer of embryos will be carry out fifth day after oocyte retrieval using a catheter.

ELIGIBILITY:
Unexplained Infertility Group; The inclusion criteria are;

1. normal HSG,
2. normal hormone levels,
3. normal over functions,
4. having normal uterine cavity and endometrial thickness determined by office hysteroscopy
5. no endometriosis (determined by transvaginal ultrasonography and / or diagnostic laparoscopy)
6. normal spermiogram result Recurrent Implantation Failure The inclusion criteria are;

1-The inclusion criteria of the working group are: 2-Failure of embryo transfer at least twice after high quality embryo transfer after 3-IVF treatment, 4-having normal hormone reserve (FSH <8 mIU / mL), 5-respond well to hormone stimulation (> 8 oocyte collection), 6-having normal uterine cavity and endometrial thickness determined by office hysteroscopy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 36 month
  Clinical pregnancy includes intrauterine gestation (pres- ence of a gestational sac on ultrasonography), ectopic preg- nancy, and miscarriage diagnosed by histology.Cycles with only a positive pregnancy test (biochemical pregnancy) are not considered to have a clinical pregnancy.
Live Birth Rate | 36 month
  A delivery is the birth of one or more infants, either living or not, after 20 weeks of gestation. A live birth is a delivery that results in at least one living infant
Abortion Rate | 36 month
  Pregnancy loss includes miscarriage and therapeutic abor- tion of a clinical intrauterine pregnancy occurring at %20 weeks of gestation.
Implantation Rate | 36 month
  Implantation rate is the number of gestational sacs observed on ultrasonog- raphy, divided by the number of embryos transferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Fulya Hospital, Istanbul, Besiktas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tasoglu S, Safaee H, Zhang X, Kingsley JL, Catalano PN, Gurkan UA, Nureddin A, Kayaalp E, Anchan RM, Maas RL, Tuzel E, Demirci U. Exhaustion of racing sperm in nature-mimicking microfluidic channels during sorting. Small. 2013 Oct 25;9(20):3374-84. doi: 10.1002/smll.201300020. Epub 2013 May 16. PMID 23677651